CLINICAL TRIAL: NCT05874648
Title: Peripheral Blood cfDNA Methylation, Fragmentation, and Proteomics for Multiple Cancers Early Detection: a Multicenter, Prospective, Observational, Case-control Study
Brief Title: PRediction Of Five Usual Tumors Using Blood Test for Risk Assessment and Early Detection
Acronym: PROFUTURE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Shanghai Weihe Medical Laboratory Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: GENIE-PROFUTURE-P
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Neoplasms; Cancer
Keywords: Cancer Screening; Blood Test; High-Throughput Nucleotide Sequencing; Circulating cell-free DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm
  Interventions: Device: Multi-cancer early detection test
- Non-cancer arm
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection test

SUMMARY:
Liquid biopsy technology based on cell-free nucleic acids and protein characteristics has unique advantages and significant application prospects in cancer early detection. The purpose of this study is to collect peripheral blood samples from participants with new diagnosis of cancer and from participants who do not have a diagnosis of cancer in order to develop machine learning models for discovering cancer from non-cancer.

DETAILED DESCRIPTION:
The PROFUTURE study: A prospective, multicenter, observational, case-control study with collection of peripheral blood and clinical data from clinical networks in order to develop machine learning models for discovering cancer from non-cancer. According to the statistical hypothesis based on expected detection performance, the study will enroll approximately 3,830 participants, including 2,138 participants with cancer (case arm) and approximately 1,692 representative participants without a clinical diagnosis of cancer after medical screening (control arm). Participants pre-matched by age and gender will be divided into training set and validation set in a ratio of approximately 7:3. The validation set will be blinded until the models are developed. Clinical information, demographics, and medical data relevant to cancer status are collected from all participants and their medical records at baseline. The participants of control arm will be asked to report suspected cancer diagnosis status within 6 months after blood collection.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* 40-75 years old
* Ability to provide a written informed consent
* Confirmed cancer diagnosis within 30 days after study blood draw, based upon assessment of a pathological specimen
* Have not received any systemic or local antitumor therapy, including but not limited to surgical resection, radiotherapy, hormone therapy, targeted therapy, immunotherapy, interventional therapy, etc.

Exclusion Criteria for Cancer Arm Participants:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Acute exacerbation of inflammatory condition or severe infection requiring therapy in hospital within 14 days prior to blood draw
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Poor health status or unfit to tolerate blood draw

Inclusion Criteria for Non-Cancer Arm Participants:

* 40-75 years old
* Ability to provide a written informed consent
* With clinically and/or pathologically diagnosed benign disease as defined by the protocol or self-reported no history of tumor and no signs of tumor as determined clinically

Exclusion Criteria for Non-Cancer Arm Participants:

* Pregnancy or lactating women
* Any tumor history of benign or malignancies
* Acute exacerbation of inflammatory condition or severe infection requiring therapy in hospital within 14 days prior to blood draw
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Poor health status or unfit to tolerate blood draw

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and communities. Participants will be assigned into two arms, including participants with new diagnosis of cancer and participants without a clinical diagnosis of cancer after medical screening. Demographic and cancer risk-related characteristics (eg, age, gender, smoking status, alcohol consumption) will be collected from all enrolled subjects.
Sampling Method: Non-Probability Sample
Enrollment: 3830 (Estimated)
Dates: Start 2023-07-07 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of predefined five types of cancers and specificity of non-cancers and in different subgroup of cfDNA methylation-based model at 95% confidence interval. | 12 months
Tissue of origin (TOO) accuracy of five types of cancers of cfDNA methylation-based model at 95% confidence interval. | 12 months

SECONDARY OUTCOMES:
Sensitivity, specificity and TOO accuracy of five types of cancers of a multi-omics model at 95% confidence interval. | 12 months
Sensitivity, specificity and TOO accuracy of cfDNA methylation-based model and multi-omics model in different stages or pathological types of five types of cancers at 95% confidence intervals. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No